CLINICAL TRIAL: NCT05149222
Title: "REACT-FM-EXT": Real-World Evidence From Smartphone-Based Acceptance and Commitment Therapy in Fibromyalgia: An Extension Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swing-003-EXT
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a virtual, single-arm, pragmatic, non-significant risk study.
  Study participants will receive 12 weeks of Digital Acceptance and Commitment Therapy (ACT) in addition to their standard care for fibromyalgia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Digital Acceptance and Commitment Therapy (ACT) Arm (Other): Pragmatic
  Interventions: Device: Digital ACT

INTERVENTIONS:
Device: Digital ACT — This is a virtual, single-arm, non-significant risk study. Study participants will receive 9 months of Digital Acceptance and Commitment Therapy (ACT) in addition to their standard care for fibromyalgia.

SUMMARY:
This is an extension study of REACT-FM. The primary objective of the study is to assess the response to digital therapy in the treatment of fibromyalgia over an additional 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed participation in the REACT-FM study.
* Participant has completed 41 sessions within Tempo in the REACT-FM study and is willing and able to comply with all protocol-specified requirements.
* Participant has provided informed consent to participate.
* Participant continues to meet original safety criteria for the REACT-FM study.

Exclusion Criteria:

* None

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the response rate to Patient Global Impression of Change (PGIC). | 9 months
  PGIC scores included are: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQ-R) total score | Enrollment to Month 9
  FIQ-R total score ranges between 0-100 with a reduction in score indicating reduced fibromyalgia severity.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) symptoms domain score | Enrollment to Month 9
  FIQ-R symptoms domain score ranges between 0-50 with a reduction in score indicating reduced fibromyalgia symptoms.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) function domain score | Enrollment to Month 9
  FIQ-R function domain score ranges between 0-30 with a reduction in score indicating improved function.
Revised Fibromyalgia Impact Questionnaire (FIQ-R) impact domain score | Enrollment to Month 9
  FIQ-R impact domain score ranges between 0-20 with a reduction in score indicating reduced fibromyalgia impact.
Participant's self-reported average weekly pain score, recorded on an NRS scale | Enrollment to Month 9
  Average pain intensity score ranges between 0-10 with a reduction in score indicating a decrease in pain intensity.
Participant's self-reported average weekly pain interference score, recorded on an NRS | Enrollment to Month 9
  Average pain interference score ranges between 0-10 with a reduction in score indicating a decrease in pain interference.
Participant's self-reported weekly sleep interference score, recorded on an NRS scale | Enrollment to Month 9
  Average sleep interference score ranges between 0-10 with a reduction in score indicating a decrease in sleep interference.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keefe, MD, Principal Investigator — Swing Therapeutics
Locations (1):
- Swing Therapeutics, San Francisco, California, United States

REFERENCES:
- See also: Swing Therapeutics Website — https://www.swingtherapeutics.com/